CLINICAL TRIAL: NCT05934812
Title: A Randomized, Placebo-controlled, Double-blind, 2-period Cross-over Study in Youth With Autism Spectrum Disorders Evaluating Social and Repetitive Behaviors After Four Weeks of Twice Daily-doses of 24IU of Intranasally Administered Oxytocin
Brief Title: Intranasal Oxytocin in Youth With Autism
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Ole A. Andreassen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-002280-10
Record Dates: First submitted 2023-06-24; First posted 2023-07-07 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): 24IU oxytocin liquid delivered with a pump-actuated nasal spray device, administered twice-daily
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator): Placebo delivered with a pump-actuated nasal spray device, administered twice-daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — 24IU oxytocin liquid delivered with a pump-actuated nasal spray device, administered twice-daily
  Arms: Oxytocin
Drug: Placebo — Placebo liquid nasal spray administered twice-daily
  Arms: Placebo

SUMMARY:
Growing evidence demonstrates the critical contribution of the neuropeptide oxytocin in the development and maintenance of autism, due to its role in social behaviour and learning processes. While some preliminary findings in oxytocin administration trials have been promising, a complete understanding of the effects of long-term oxytocin administration in autism remains elusive, as participant numbers in oxytocin administration studies in autism have been small, most studies exclusively recruit males, and reproducibility has been inconsistent.

To address this critical knowledge gap, this project will include a double-blind, placebo-controlled, randomized controlled crossover trial of a four-week intranasal oxytocin treatment (24 international units, twice-daily) in 128 male and female youth with ASD aged 12-20, with social and repetitive behaviors as primary outcome measures. The investigators predict that intranasal oxytocin treatments will increase performance on social behavior measures and reduce repetitive behaviors using caregiver-reported measures.

Along with the investigation of oxytocin's long-term effects, the investigators will also assess the impact of oxytocin administration on computer-based laboratory tasks that can precisely measure how participants process social cues and disengage with repetitive behaviours. In addition, an electrocardiogram will be collected to evaluate the impact of oxytocin administration on parasympathetic nervous system activity.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants between the ages of 12 and 20, both inclusive, with a confirmed diagnosis of autism spectrum disorder (ASD) diagnosis as per the ADOS/ADI.
2. Participants must be in good general physical health, as determined by the investigator.
3. Participant's pre-study physical examination and vital signs must not show any clinically significant abnormalities as determined by the investigator.
4. Participants and caregivers must be able to communicate well with the investigator, to understand and comply with the requirements of the study, and to understand the oral and written study information

Exclusion Criteria:

1. Previous nasal disease, surgery, and dependence on inhaled drugs.
2. Current significant nasal congestion due to common colds.
3. Clinically relevant history of significant hepatic, renal, endocrine, cardiac, nervous, pulmonary, haematological or metabolic disorder.
4. Systemic illness requiring treatment within 2 weeks prior to Study Day 1.
5. Full scale IQ < 70 (due to the prerequisite ability to complete self-report measures).
6. Known allergic reactions or hypersensitivity to any component of the study medication in the nasal spray, such as propyl parahydroxybenzoate (E216), methyl parahydroxybenzoate (E218) and chlorobutanol hemihydrate.
7. Known allergic reactions or hypersensitivity/intolerance to latex
8. Currently breastfeeding
9. Pregnancy (self-reported or assessed by pregnancy test prior to the first administration at Experimental session 1 and 2 for all menstruating females)
10. Participation in any (other) clinical trial with an investigational medicinal product or medical device within 3 months prior to randomisation.
11. New concomitant medications or formal cognitive/behavioral therapies. If a participant has been taking any medications or receiving formal cognitive/behavioral therapies for at least 4 weeks, then this is not considered a new therapy.
12. Other unspecified reasons that, in the opinion of the investigator or the sponsor make the participants unsuitable for enrolment.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-09-18 (Estimated); Primary Completion 2025-11-04 (Estimated); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
Social behavior | Four weeks
  Assessed by the total score of the Social Responsiveness Scale-Second Edition (SRS-2), as completed by caregivers of the participants. Lower scores represent better outcomes.
Repetitive behaviour | Four weeks
  Assessed with the Repetitive Behavior Scale-Revised (RBS-R), as completed by caregivers of the participants. Lower scores represent better outcomes.

SECONDARY OUTCOMES:
Behavioral inflexibility | Four weeks
  Assessed by the Behavioral inflexibility scale (BIS), completed by caregivers of the participants. Lower scores represent better outcomes.
Social cognition | Four weeks
  Assessed by a computerized Emotional body language task completed by the participants. Higher accuracy scores represent better outcomes.
Repetitive cognition | Four weeks
  Assessed by a computerised probabilistic reversal learning task completed by participants. More regressive errors represent worse outcomes (i.e., after initially choosing the new correct response, participants regress back to choosing the previously rewarded response)
Vagally-mediated heart rate variability | Four weeks
  Calculated using electrocardiogram (RMSSD and High Frequency HRV)

OTHER OUTCOMES:
Participation in social activities | Four weeks
  As measured by the Participation and Environment measure-Child and Youth scale. Higher scores on the "participation frequency", "level of involvement", and "Percent total environmental supportiveness" subscores represent better outcomes, and lower scores on the "Percent never participates" and "Percent that parents desired change" represent better outcomes
Caregiver quality of life | Four weeks
  As measured by the Care-related Quality of Life instrument (CarerQol). Higher scores represent better outcomes
Executive function | Four weeks
  As measured by the Behavior Rating Inventory of Executive Functions. Lower scores represent better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ole A Andreassen, PhD, MD, Principal Investigator — University of Oslo
Locations (1):
- Ullevål Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
This needs to confirmed with local data protection authorities